CLINICAL TRIAL: NCT07000175
Title: Comparison of Heart Rate Variability Measurement on the Arm and Chest in Transcutaneous Auricular Vagus Nerve Stimulation
Brief Title: Comparison of Heart Rate Variability Measurement on the Arm and Chest in Vagus Nerve Stimulation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, Alper Percin, Asst. Prof., Bahçeşehir University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: AVU10002
Record Dates: First submitted 2025-05-23; First posted 2025-06-02 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Sympathetic; Imbalance
Keywords: Heart Rates; Vagus Nerves

STUDY DESIGN:
Intervention Model Description: A modelling will be created in which the same intervention will be applied to the three groups but the evaluations will be made differently.
Who Masked: Investigator
Masking Description: Single blinding (investigator blinding)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Measurement over the chest (Active Comparator): Heart rate variability will be measured on the chest for 5 minutes before and after transcutaneous vagus nerve stimulation.
  Interventions: Device: Transcutaneous Auricular Vagus Nerve Stimulation
- Measurement over the right arm (Active Comparator): Heart rate variability will be measured on the right arm for 5 minutes before and after transcutaneous vagus nerve stimulation.
  Interventions: Device: Transcutaneous Auricular Vagus Nerve Stimulation
- Measurement over the left arm (Active Comparator): Heart rate variability will be measured on the left arm for 5 minutes before and after transcutaneous vagus nerve stimulation.
  Interventions: Device: Transcutaneous Auricular Vagus Nerve Stimulation

INTERVENTIONS:
Device: Transcutaneous Auricular Vagus Nerve Stimulation — Non-invasive transcutaneous vagus nerve stimulation with special earphones placed in the ear will be applied to the participants for 20 minutes and a single session.

SUMMARY:
Healthy participants will be included in this study by invitation and randomised into three groups. Participants in each group will receive bilateral transcutaneous vagus nerve stimulation with the same frequency, current transit time and current intensity. Heart rate variability will be measured over the chest in the first group, over the right arm in the second group and over the left arm in the third group. Then, the differences between the groups in heart rate variability parameters (time-dependent, frequency-dependent) will be compared. The aim of this study is to examine the differences between heart rate variability measurements measured at different sites.

DETAILED DESCRIPTION:
Heart rate variability is defined as the change in beat-to-beat interval, and the sympathetic and parasympathetic nervous system influences the change in beat-to-beat interval through cardiovascular connections. Heart rate variability measurement can be obtained by different methods. However, which method is more effective is controversial. The aim of this study was to investigate the differences between heart rate variability parameters measured on the chest, right arm and left arm.

Healthy participants aged 18-45 years will be included in the study. The inclusion criteria will be determined as being 18 years of age or older and not having any acute or chronic disease. Exclusion criteria will be determined as being previously involved in any neuromodulation intervention, smoking or alcohol use, and regular medication use.

Participants included in the study will be randomised into three groups and transcutaneous vagus nerve stimulation will be applied. The duration of treatment will be 20 minutes and single session stimulation will be performed. Current intensity, current passage time and frequency will be planned to be the same in each patient. Before and after stimulation, heart rate variability will be measured over the chest in the first group, over the right arm in the second group and over the left arm in the third group. Then, heart rate variability parameters (time-dependent, frequency-dependent) will be compared between the groups.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* To know how to read and write Turkish
* Not having any acute or chronic disease

Exclusion Criteria:

* Previous application of any neuromodulation method
* Smoking or alcohol use
* Use of any supplementary medication

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Estimated)
Dates: Start 2025-05-30 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Heart Rate Variability | Baseline and after 20 minutes of treatment
  Heart rate variability will be measured with a 5-minute short measurement method over the chest, right arm and left arm.

CONTACTS AND LOCATIONS:
Overall Officials: Ramazan Cihad Yılmaz, Ph.D., Study Director — Igdir University
Locations (1):
- Avrasya University Physical Therapy Laboratory, Trabzon, Ortahisar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gillinov S, Etiwy M, Wang R, Blackburn G, Phelan D, Gillinov AM, Houghtaling P, Javadikasgari H, Desai MY. Variable Accuracy of Wearable Heart Rate Monitors during Aerobic Exercise. Med Sci Sports Exerc. 2017 Aug;49(8):1697-1703. doi: 10.1249/MSS.0000000000001284. PMID 28709155